CLINICAL TRIAL: NCT03540030
Title: Opioid-Free Shoulder Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00021833
Record Dates: First submitted 2018-05-08; First posted 2018-05-30 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Opioid Use; Shoulder Osteoarthritis; Avascular Necrosis; Rotator Cuff Tear; Arthritis;Inflammatory
Keywords: Primary Total Shoulder Arthroplasty; Reverse Total Shoulder Arthroplasty
MeSH Terms: conditions — Osteonecrosis; Rotator Cuff Injuries; Arthritis | interventions — Gabapentin; Celecoxib; Ketorolac Tromethamine; Acetaminophen; Propofol; Lidocaine; Rocuronium; Vecuronium Bromide; Sevoflurane; Desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Observational (No Intervention): The observational treatment group will not have any changes from your surgeon's normal pain management process. Anesthesia will be utilized in a routine fashion with all routine perioperative medications. You will be discharged on routine postoperative medications including opioids, NSAIDS, and any other modalities typically used by the treating surgeon.
- Non-Opioid Intervention (Active Comparator): Oral dose of both gabapentin and celecoxib (toradol if sulfa allergy) in the preop area. US-guided interscalene regional block without the aid of opioid co-medication. Intra-op management by anesthesia with non-opioid modalities but should include one dose of IV acetaminophen during the procedure. Anesthetic modalities will include, but not limited to, regional block, propofol, IV lidocaine, rocuronium/vecuronium, and sevoflurane/desflurane. If the attending anesthesiologist deems it necessary to dose with opioids during procedure, it will be recorded and reported. Liposomal bupivacaine will be injected into the peri-articular soft tissues as an adjunct to the block. Post Op, cryotherapy, gabapentin, toradol. Toradol will transition to celecoxib for the duration of the hospitalization (or meloxicam for patients with sulfa allergy). As needed medications will include both oral and IV acetaminophen, as well as up to an additional 15mg of toradol per 6hr, depending on Cr clearance.
  Interventions: Drug: Gabapentin; Drug: Celecoxib; Drug: toradol; Drug: acetaminophen; Drug: regional block; Drug: propofol; Drug: IV lidocaine; Drug: rocuronium; Drug: vecuronium; Drug: sevoflurane; Drug: desflurane

INTERVENTIONS:
Drug: Gabapentin — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: Celecoxib — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: toradol — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: acetaminophen — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: regional block — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: propofol — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: IV lidocaine — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: rocuronium — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: vecuronium — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: sevoflurane — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention
Drug: desflurane — opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment
  Arms: Non-Opioid Intervention

SUMMARY:
Purpose of Study:

To identify and provide a safe, opioid-free treatment pathway for shoulder arthroplasty with a focus on perioperative pain control and postoperative symptoms from treatment

DETAILED DESCRIPTION:
Background and Significance:

Opioid-based analgesia has been a cornerstone of patient care in the setting of acute pain for the last century and has undergone logarithmic increase over the past twenty years. Unfortunately, the rise in utilization has brought with it a rise in opioid-induced side effects. These include constipation, nausea/vomiting, hyperalgesia, delirium, addiction/withdrawal (with 67% of those prescribed a long-term opioid program still on opioids at an average of 4.8 years of follow-up), and in some cases even respiratory depression/death. Patient expectations of opioid-based pain medication has driven a rapid rise in outpatient opioid prescriptions including both short and long-acting opioids. These prescriptions have in turn become a source of significant mortality in the United States, with nearly 20,000 deaths due to opioid overdose in 2014 alone.

There have been momentous efforts made in identifying synergistic compounds to use for acute pain management in the perioperative time period to begin to minimize the opioid requirement for pain control. These studies have focused on nerve modulation with gabapentinoids, intravenous and local administration of sodium-channel blockers such as lidocaine and bupivacaine, and even increased interest in non-steroidal anti-inflammatories and acetaminophen. At this time, no study has looked at the possibility of utilizing a multi-modal acute post-surgical pain control pathway that did not include some form of opioid medication for the general population.

Arthroplasty continues to be a dominant procedure in the orthopaedic armamentarium and accounts for well over a million surgeries done in the United States per year. With the ability to utilize targeted nerve blocks by anesthesia, and the increasing data showing efficacy of multi-modal therapy for acute pain, we propose a patient care pathway that is completely free of all opioid-based medications. From the time that patients are checked in until the time the patient follows up in clinic, they will utilize a pathway designed to eliminate pain and opioid-related side effects following shoulder arthroplasty. Our hope is that a well-designed pathway for total shoulder arthroplasty can quickly be modeled for other surgical procedures in an attempt to minimize the negative effects of opioid utilization both acutely and on a societal level.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing elective primary total shoulder or reverse total shoulder arthroplasty for osteoarthritis, avascular necrosis, cuff tear arthropathy, or inflammatory arthritis etiologies
2. Age greater than or equal to 50.

Exclusion Criteria:

1. Revision total shoulder arthroplasty
2. Chronic opioid therapy - per investigator discretion
3. Liver or renal insufficiency - per investigator discretion
4. Arthroplasty for fracture
5. Sickle cell disease
6. Workers compensation
7. Inability to receive block
8. Intervention Arm Only: Creatinine clearance less than 30 mL/min
9. Intervention Arm Only: Allergy to non-steroidal anti-inflammatory medications (NSAIDs).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoCarolina Research Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Lee HJ, Yeomans DC. Opioid induced hyperalgesia in anesthetic settings. Korean J Anesthesiol. 2014 Nov;67(5):299-304. doi: 10.4097/kjae.2014.67.5.299. Epub 2014 Nov 26. PMID 25473457
- [Background] McKeown JL. Pain Management Issues for the Geriatric Surgical Patient. Anesthesiol Clin. 2015 Sep;33(3):563-76. doi: 10.1016/j.anclin.2015.05.010. Epub 2015 Jul 3. PMID 26315638
- [Background] Macintyre PE, Huxtable CA, Flint SL, Dobbin MD. Costs and consequences: a review of discharge opioid prescribing for ongoing management of acute pain. Anaesth Intensive Care. 2014 Sep;42(5):558-74. doi: 10.1177/0310057X1404200504. PMID 25233168
- [Background] Seib RK, Paul JE. Preoperative gabapentin for postoperative analgesia: a meta-analysis. Can J Anaesth. 2006 May;53(5):461-9. doi: 10.1007/BF03022618. PMID 16636030
- [Background] Doleman B, Heinink TP, Read DJ, Faleiro RJ, Lund JN, Williams JP. A systematic review and meta-regression analysis of prophylactic gabapentin for postoperative pain. Anaesthesia. 2015 Oct;70(10):1186-204. doi: 10.1111/anae.13179. Epub 2015 Aug 24. PMID 26300519
- [Background] Mishriky BM, Waldron NH, Habib AS. Impact of pregabalin on acute and persistent postoperative pain: a systematic review and meta-analysis. Br J Anaesth. 2015 Jan;114(1):10-31. doi: 10.1093/bja/aeu293. Epub 2014 Sep 10. PMID 25209095
- [Background] Banerjee P, Rogers BA. Systematic review of high-volume multimodal wound infiltration in total knee arthroplasty. Orthopedics. 2014 Jun;37(6):403-12. doi: 10.3928/01477447-20140528-07. PMID 24972430
- [Background] Marques EM, Jones HE, Elvers KT, Pyke M, Blom AW, Beswick AD. Local anaesthetic infiltration for peri-operative pain control in total hip and knee replacement: systematic review and meta-analyses of short- and long-term effectiveness. BMC Musculoskelet Disord. 2014 Jul 5;15:220. doi: 10.1186/1471-2474-15-220. PMID 24996539
- [Background] Skolnik A, Gan TJ. New formulations of bupivacaine for the treatment of postoperative pain: liposomal bupivacaine and SABER-Bupivacaine. Expert Opin Pharmacother. 2014 Aug;15(11):1535-42. doi: 10.1517/14656566.2014.930436. Epub 2014 Jul 3. PMID 24992382
- [Background] Kazerooni R, Tran MH. Evaluation of Celecoxib Addition to Pain Protocol After Total Hip and Knee Arthroplasty Stratified by Opioid Tolerance. Clin J Pain. 2015 Oct;31(10):903-8. doi: 10.1097/AJP.0000000000000178. PMID 25380221
- [Background] Khan JS, Margarido C, Devereaux PJ, Clarke H, McLellan A, Choi S. Preoperative celecoxib in noncardiac surgery: A systematic review and meta-analysis of randomised controlled trials. Eur J Anaesthesiol. 2016 Mar;33(3):204-14. doi: 10.1097/EJA.0000000000000346. PMID 26760402
- [Background] Koh W, Nguyen KP, Jahr JS. Intravenous non-opioid analgesia for peri- and postoperative pain management: a scientific review of intravenous acetaminophen and ibuprofen. Korean J Anesthesiol. 2015 Feb;68(1):3-12. doi: 10.4097/kjae.2015.68.1.3. Epub 2015 Jan 28. PMID 25664148
- [Background] Nir RR, Nahman-Averbuch H, Moont R, Sprecher E, Yarnitsky D. Preoperative preemptive drug administration for acute postoperative pain: A systematic review and meta-analysis. Eur J Pain. 2016 Aug;20(7):1025-43. doi: 10.1002/ejp.842. Epub 2016 Mar 15. PMID 26991963
- [Background] Rouhani A, Tabrizi A, Elmi A, Abedini N, Mirza Tolouei F. Effects of preoperative non-steroidal anti-inflammatory drugs on pain mitigation and patients' shoulder performance following rotator cuff repair. Adv Pharm Bull. 2014 Dec;4(4):363-7. doi: 10.5681/apb.2014.053. Epub 2014 Aug 10. PMID 25436192
- [Background] Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the Real Benefits of Single-Shot Interscalene Block Please Stand Up? A Systematic Review and Meta-Analysis. Anesth Analg. 2015 May;120(5):1114-1129. doi: 10.1213/ANE.0000000000000688. PMID 25822923
- [Background] Chan EY, Fransen M, Parker DA, Assam PN, Chua N. Femoral nerve blocks for acute postoperative pain after knee replacement surgery. Cochrane Database Syst Rev. 2014 May 13;2014(5):CD009941. doi: 10.1002/14651858.CD009941.pub2. PMID 24825360
- [Background] Ullah H, Samad K, Khan FA. Continuous interscalene brachial plexus block versus parenteral analgesia for postoperative pain relief after major shoulder surgery. Cochrane Database Syst Rev. 2014 Feb 4;2014(2):CD007080. doi: 10.1002/14651858.CD007080.pub2. PMID 24492959
- [Background] Aasvang EK, Luna IE, Kehlet H. Challenges in postdischarge function and recovery: the case of fast-track hip and knee arthroplasty. Br J Anaesth. 2015 Dec;115(6):861-6. doi: 10.1093/bja/aev257. Epub 2015 Jul 25. PMID 26209853
- [Background] Dahl JB, Nielsen RV, Wetterslev J, Nikolajsen L, Hamunen K, Kontinen VK, Hansen MS, Kjer JJ, Mathiesen O; Scandinavian Postoperative Pain Alliance (ScaPAlli). Post-operative analgesic effects of paracetamol, NSAIDs, glucocorticoids, gabapentinoids and their combinations: a topical review. Acta Anaesthesiol Scand. 2014 Nov;58(10):1165-81. doi: 10.1111/aas.12382. Epub 2014 Aug 14. PMID 25124340
- [Background] Dunn LK, Durieux ME, Nemergut EC. Non-opioid analgesics: Novel approaches to perioperative analgesia for major spine surgery. Best Pract Res Clin Anaesthesiol. 2016 Mar;30(1):79-89. doi: 10.1016/j.bpa.2015.11.002. Epub 2015 Nov 24. PMID 27036605
- [Background] Halawi MJ, Grant SA, Bolognesi MP. Multimodal Analgesia for Total Joint Arthroplasty. Orthopedics. 2015 Jul 1;38(7):e616-25. doi: 10.3928/01477447-20150701-61. PMID 26186325
- [Background] Hojer Karlsen AP, Geisler A, Petersen PL, Mathiesen O, Dahl JB. Postoperative pain treatment after total hip arthroplasty: a systematic review. Pain. 2015 Jan;156(1):8-30. doi: 10.1016/j.pain.0000000000000003. PMID 25599296
- [Background] McCartney CJ, Nelligan K. Postoperative pain management after total knee arthroplasty in elderly patients: treatment options. Drugs Aging. 2014 Feb;31(2):83-91. doi: 10.1007/s40266-013-0148-y. PMID 24399578
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] YaDeau JT, Gordon MA, Goytizolo EA, Lin Y, Fields KG, Goon AK, Holck G, Miu TW, Gulotta LV, Dines DM, Craig EV. Buprenorphine, Clonidine, Dexamethasone, and Ropivacaine for Interscalene Nerve Blockade: A Prospective, Randomized, Blinded, Ropivacaine Dose-Response Study. Pain Med. 2016 May;17(5):940-60. doi: 10.1093/pm/pnv010. Epub 2015 Dec 14. PMID 26814246
- [Background] Michener LA, Snyder AR, Leggin BG. Responsiveness of the numeric pain rating scale in patients with shoulder pain and the effect of surgical status. J Sport Rehabil. 2011 Feb;20(1):115-28. doi: 10.1123/jsr.20.1.115. PMID 21411827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were identified in clinic by the surgeon performing the shoulder arthroplasty. The surgeon introduced the concept of opioid-free arthroplasty with the patients, who then chose whether to follow the traditional or opioid-free pathway. The surgeon then notified the study coordinator of the patient's decision and patients were consented.
Groups:
- Non-Opioid Intervention: Oral dose of gabapentin and celecoxib (toradol if sulfa allergy) in the preop area. US-guided interscalene regional block without aid of opioid co-medication. Intra-op management by anesthesia with non-opioid modalities but included one dose of IV acetaminophen during procedure. Anesthetic modalities include, but not limited to, regional block, propofol, IV lidocaine, rocuronium/vecuronium, and sevoflurane/desflurane. If the attending anesthesiologist deems it necessary to dose with opioids during procedure, it will be recorded and reported. Liposomal bupivacaine will be injected into the peri-articular soft tissues as an adjunct to the block. Post Op, cryotherapy, gabapentin, toradol. Toradol will transition to celecoxib for the duration of the hospitalization (or meloxicam for patients with sulfa allergy). PRN medications will include acetaminophen, as well as up to an additional 15mg of toradol per 6hr, depending on Cr clearance.
Period: Overall Study
Arm/Group | Observational | Non-Opioid Intervention
Started | 48 | 38
Completed | 30 | 35
Not Completed | 18 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — screen fail | 7 | 1
Not completed — never had surgery after signing consent | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observational | Non-Opioid Intervention | Total
Number analyzed (Participants) | 30 | 35 | 65
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72.5 [66.3 to 78.4] | 71.1 [68.5 to 73.3] | 72.0 [66.9 to 74.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 10 | 17 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 35 | 65

OUTCOME MEASURES:

1. Primary Outcome: Post Op Pain
Description: Pain at patient discharge or 24-hours, whichever comes first - measured on a 0 (no pain) -10 (worst possible pain) numeric rating scale (NRS). A score of 0(no pain) is preferable to 10(worst possible pain)
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
score on a scale | 3.0 [1 to 5] | 2.0 [0 to 5]
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = .297, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Additional Post Op Pain
Description: post-operative pain: measured on a 0 (no pain) -10 (worst) numeric rating scale (NRS) at 6hrs, 12hrs, 2 weeks, and 2 months. A score of 0(no pain) is preferable to 10(worst possible pain)
Time Frame: 6hrs, 12hrs, 2weeks, 2 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
score on a scale
  6 Hrs | 2 [0 to 3.5] | 0.0 [0 to 0]
  12 hrs | 4 [1 to 7] | 0 [0 to 3]
  2 weeks | 1.3 [0 to 4.6] | 0.82 [0 to 3]
  2 months | 0.7 [0 to 2.9] | 0 [0 to 1.4]
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney) — At the 6 hour time point
Statistical Analysis 2: Comparison: Observational vs Non-Opioid Intervention; At the 12 hour time point; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Nausea
Description: rate of nausea
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Participants
  Yes | 5 | 1
  No | 23 | 34
  Unknown | 2 | 0
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = 0.0801, Fisher Exact

4. Secondary Outcome: Constipation
Description: rate of constipation
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Participants
  Yes | 19 | 13
  No | 9 | 22
  Unknown | 2 | 0
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = 0.0154, Chi-squared

5. Secondary Outcome: Falls
Description: rate of falls
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Participants
  Yes | 1 | 5
  No | 27 | 30
  Unknown | 2 | 0
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = 0.2139, Fisher Exact

6. Secondary Outcome: Morphine Use
Description: Morphine milli-equivalents In-hospital post-operative. Continuous scale of MME, no defined better/worse. Measured as number and dose of medications taken. For example, if the patient received an opioid, the drug and dose was recorded and converted to MME. A time frame of when to assess opioid use in-hospital post-operative was not used but was a continuous monitor for rescue opioid from in-hospital post-operative through discharge.
Time Frame: In-hospital Stay
Measure: Median (Inter-Quartile Range); unit: Morphine milli-equivalents
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Morphine milli-equivalents | 45.0 [34.0 to 66.0] | 19.0 [19.0 to 19.0]

7. Secondary Outcome: Pain Satisfaction
Description: Satisfaction with overall pain using Numeric Pain Rating (NRS) scale. yes, no. No being better than yes.
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Participants
  Yes | 27 | 34
  No | 1 | 1
  Unknown | 2 | 0
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p > .99, Fisher Exact

8. Secondary Outcome: ASES
Description: American Shoulder and Elbow Surgeons (ASES) Shoulder Score for pain and function. Range 0-100. Low score = worse shoulder condition. Function, disability, and pain subscores (all ranges 0-50), and are summed for total ASES score.
Time Frame: 2 Weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
units on a scale | 54.3 [50.2 to 62.9] | 54.2 [46.7 to 60.0]
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = 0.9669, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Simple Shoulder Test
Description: Simple Shoulder Test (SST) activity score. Range 0-12. 0 = worse activity score.
Time Frame: 2 Weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
score on a scale | 2.0 [1.5 to 4.0] | 2.0 [1.0 to 4.0]
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = .9208, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Veterans RAND 12 Item Health Survey (VR-12©) Physical Health Subscore, and Mental Health Subscore
Description: quality of life using VR-12 subscores. Physical Health (PCS) subscore and Mental Health (MCS) subscore, not summed. Range reported in weighted units. Physical Health subscore: 1 point increase in PCS is associated with 6% lower total health care expenditures, 5% lower pharmacy expenditures, 9% lower rate of hospital inpatient visits, 4% lower rate of medical provider visits, 5% lower rate of hospital outpatient visits. Mental Health sub score a 1 point increase in MCS is associated with 7% lower total health care expenditures, 4% lower pharmacy expenditures, 15% lower rate of hospital inpatient visits, and 4% lower rate of medical provider visits. Both PCS/MCS are score 0-100 with 100 indicating the highest level of health.
Time Frame: 2 Weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
score on a scale
  PCS | 36.7 [28.3 to 43.9] | 35.0 [29.1 to 43.7]
  MCS | 56.3 [50.2 to 62.9] | 59.1 [52.5 to 64.1]
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; For PCS only; Test type: Other; p = 0.6481, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Observational vs Non-Opioid Intervention; For MCS only; Test type: Other; p = 0.3911, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Nausea
Description: rate of nausea
Time Frame: 2 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Participants
  Yes | 0 | 1
  No | 28 | 30
  Unknown | 2 | 0
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p > .99, Fisher Exact

12. Secondary Outcome: Constipation
Description: rate of constipation
Time Frame: 2 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Participants
  Yes | 7 | 4
  No | 21 | 27
  Unknown | 2 | 4
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = 0.3177, Fisher Exact

13. Secondary Outcome: Falls
Description: rate of falls
Time Frame: 2 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Participants
  Yes | 4 | 4
  No | 24 | 27
  Unknown | 2 | 4
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p > .99, Fisher Exact

14. Secondary Outcome: Pain Satisfaction
Description: Satisfaction with overall pain using Numeric Pain Rating (NRS) scale. yes, no. No being better than yes.
Time Frame: 2 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
Participants
  Yes | 23 | 29
  No | 5 | 2
  Unknown | 2 | 4
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = 0.2349, Fisher Exact

15. Secondary Outcome: Simple Shoulder Test
Description: Simple Shoulder Test (SST) activity score. Range 0-12. 0 = worse activity score.
Time Frame: 2 Months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
score on a scale | 6 [4 to 9] | 6 [4 to 7]
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; Test type: Other; p = 0.7892, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Veterans RAND 12 Item Health Survey (VR-12©) Physical Health Subscore, and Mental Health Subscore
Description: as for outcome 10
Time Frame: 2 Months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Observational | Non-Opioid Intervention
Number analyzed (Participants) | 30 | 35
score on a scale
  PCS | 38.4 [29.6 to 44.9] | 40.3 [33.8 to 47.0]
  MCS | 58.7 [47.6 to 62.7] | 60.8 [49.4 to 64.0]
Statistical Analysis 1: Comparison: Observational vs Non-Opioid Intervention; For PCS only; Test type: Other; p = 0.2023, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Observational vs Non-Opioid Intervention; For MCS only; Test type: Other; p = 0.2486, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of study treatment (surgery) through the end of subject participation (1 year postoperative visit).
Arm/Group | Observational | Non-Opioid Intervention
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/48 | 2/38
Other Adverse Events (participants affected / at risk) | 0/48 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational (N=48) | Non-Opioid Intervention (N=38)
Hospitalization for ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient was hospitalized for >24 hours for an ileus. Determined to be not related to the study.
DVT and pulmonary embolism (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Patient was hospitalized for >24 hours for a deep vein thrombosis and pulmonary embolism. Determined to be unlikely related to the study.
mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Patient was hospitalized >24 hours for lower quadrant abdominal pain diagnosed as mesenteric artery stenosis. Determined to be unlikely related to study.

LIMITATIONS AND CAVEATS:
Enrollment into either pathway was voluntary, not randomized. Patient-kept diaries are difficult data to rely on. Only examines the short-term recovery of the patients undergoing TSA/RTSA. Did not evaluate the cost with each treatment arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03540030/Prot_SAP_000.pdf